CLINICAL TRIAL: NCT05766917
Title: Effectiveness of Peer Education on Core Health Outcomes Specific for Burn Patients: Randomized Controlled Study
Brief Title: Peer Education on Core Health Outcomes Specific for Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Heba Abubakr Mohamed Salama, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Peer education burn patients
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Burns
Keywords: Burn Specific Health Scale; Burn patients; Peer education
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): this group will receive the routine hospital care provided in burn center
- peer education group (Experimental): this group will receive the routine hospital care, in addition to the proposed peer education by trained peer.
  Interventions: Behavioral: peer education group

INTERVENTIONS:
Behavioral: peer education group — Patients in this group will receive the routine hospital care, in addition to the proposed peer education by trained peer
  Arms: peer education group

SUMMARY:
Evaluate the Effectiveness of Peer Education on Core Health Outcomes Specific for Burn Patients

DETAILED DESCRIPTION:
A randomized controlled study will done in the Plastic & Reconstructive Burn Center at Mansoura University Hospitals. the first phase includes the systematic collection of data to assess patient's health status and determine any actual or potential health problems after necessary permission taken.

The researcher will design the proposed peer education and educational media based on the findings of the assessment.

After peers training, implementing peer education for the study group. The final step of data collection is evaluating the patient's response to the proposed program and the extent to which the outcomes have been achieved.

ELIGIBILITY:
Inclusion Criteria for patients:

Recently admitted patients

* Hemodynamically stable and Free from chronic disease
* Conscious, able to communicate

Inclusion criteria for peer:

* old burns injury patients at least have a diploma degree

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
change in Burn Specific Health Scale measurements | 3 months
  the outcome will be measured three times (before , after intervention and after three months ) The scoring system will performed as follows: responses to each of the 40 items are rated on a five- point scale from zero (extremely) to four (not at all) for each of the 40 items. Mean scores are calculated for each domain. The maximum score was 160 points and the minimum score was 0. A higher mean score indicates more positive evaluation of patients core health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ola E Elsherbiny, pHD, Study Chair — Mansoura University, Faculty of Nursing
Locations (1):
- Heba Abubakr Salama, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No